CLINICAL TRIAL: NCT01724684
Title: Feasibility and Effectiveness of Telehealth in Patients With Chronic Obstructive Pulmonary Disease in Taiwan
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 201106097RB
Record Dates: First submitted 2012-01-02; First posted 2012-11-12 (Estimated); Last update posted 2012-11-12 (Estimated); Status verified 2012-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telehealth program (Other): Telehealth program service
  Interventions: Other: Telehealth program
- Usual care (Other): Usual care service
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Telehealth program
  Arms: Telehealth program
Other: Usual care
  Arms: Usual care

SUMMARY:
Recent studies have demonstrated the promising potential that telehealth has in management of chronic disease. For COPD patients, implementation of telehealth reduced readmissions, emergency room visits, and exacerbations and was cost-effective. Telehealth as a method of delivering healthcare to remote, resource-deprived areas is not lacking in evidence of benefit; however, the situation about its more widespread use for monitoring purposes is much less clear. To date, most of the studies dealing with telehealth in COPD were conducted in countries covering vast territories. Therefore, it needs to be investigated whether telehealth conveys similar advantages for COPD patients in a small island country.

ELIGIBILITY:
Inclusion Criteria:

* Admissions for chronic obstructive pulmonary disease
* Age 20 or more

Exclusion Criteria:

* Discharge against medical advice
* Enrolled in other trials
* Not being discharged to home
* Unconsciousness

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-12; Primary Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Hospital Readmission at 6 months | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Ta Huang, M.D, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan

REFERENCES:
- [Derived] Cox NS, Dal Corso S, Hansen H, McDonald CF, Hill CJ, Zanaboni P, Alison JA, O'Halloran P, Macdonald H, Holland AE. Telerehabilitation for chronic respiratory disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013040. doi: 10.1002/14651858.CD013040.pub2. PMID 33511633